CLINICAL TRIAL: NCT00840931
Title: A Phase I Pilot Study of Immunotherapy Using Lenalidomide Plus "Bystander" Vaccine in Patients With High-Risk Myelodysplastic Syndrome (MDS)
Brief Title: Immunotherapy Using Lenalidomide + Bystander Vaccine in High Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14998; 105861 (Other: USF IRB); RV-MDS-PI-202 (Other: Celgene Corp.); BB-IND 13478 (Other: CBER); 0803-907 (Other: OBA)
Record Dates: First submitted 2009-02-04; First posted 2009-02-11 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Leukemia
Keywords: Myeloid; Monocytic; Immunotherapy; Vaccine; MDS; High Risk Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immunotherapy (Experimental): Participants will take two 5 mg capsules of lenalidomide per day for 21 days followed by 7 days of rest. This 28 day period is considered 1 cycle. Participants will receive 4 treatment cycles with 28 days in each cycle. Those participants showing a clinical response after 4 cycles of treatment may continue to receive lenalidomide as a single agent for additional cycles at the treating Physicians discretion. During each 28 day cycle participants will also receive GM.CD40L bystander vaccination injections in 2-week intervals on days 8 and 22 for a total of 8 immunizations during the 4 cycle treatment period.
  Interventions: Drug: lenalidomide; Biological: bystander vaccine

INTERVENTIONS:
Drug: lenalidomide — Patients will take 10 mg capsules of lenalidomide per day for 21 days followed by 7 days of rest. This 28 day period is considered 1 cycle. Patients will receive 4 treatment cycles with 28 days in each cycle.
  Other Names: Revlimid®
Biological: bystander vaccine — In addition to lenalidomide, during each 28 day cycle patients will also receive GM.CD40L bystander vaccination injections in 2-week intervals on days 8 and 22 for a total of 8 immunizations during the 4 cycle treatment period.
  Other Names: GM.CD40L

SUMMARY:
The purpose of this study is to find out the maximum tolerated dose (MTD) of the combined therapy of lenalidomide (Revlimid®) and Granulocyte/macrophage colony stimulating factor and CD40 Ligand expressed in the K562 cell line (GM.CD40L) bystander vaccine. This research is also being done to see how well the combination of these drugs works to fight myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
Fixed dose of lenalidomide at 10 mg/day, Days 1- 21 of 28 days of treatment cycle, and 4 dose escalations of GM.CD40L vaccine: 10 X 10^6 GM.CDL cells per vaccination; 30 X 10^6 GM.CDL cells per vaccination; 60 X 10^6 GM.CDL cells per vaccination; 120 X 10^6 GM.CDL cells per vaccination; Vaccination at 2-week intervals, on days 8 and 22, for a total of four 28-day cycles.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form
* Age ≥18 years at the time of signing the informed consent form
* Able to comply with the study visit schedule and assessments required by the protocol
* Documented diagnosis of MDS with subtypes of Refractory Anemia with Excess Blast 1 (RAEB-1) (myeloblast ≥5-9%) or Refractory Anemia with Excess Blast 2 (RAEB-2) (myeloblast ≥10-19%) or intermediate 2, Acute myelogenous leukemia with bone marrow myeloblast >30% and high risk defined by International Prognostic Scoring System (IPSS) scores or refractory anemia with excess blast in transformation (RAEB-t) (myeloblast ≥ 20-30%) as per French-American-British Classification System (FAB) criteria. Any single or combination of cytogenetic abnormalities is allowed.
* Study treatment can be offered as first line treatment as long as the available food and Drug Administration (FDA) approved treatment options are explained by the treating physician and the participant declines such options.
* Study treatment can be offered to patients who have failed, cannot tolerate or do not wish to continue other therapeutic agents for MDS.
* Prior chemotherapy is allowed but should be off chemotherapy of any kind for at last 4 weeks prior to initiation of study therapy.
* Must be able to provide adequate bone marrow (BM) aspirate and biopsy specimens for histopathological evaluation, cytogenetic analysis and tissue banking during the screening procedure.
* Platelet count must be > 20,000/ µl without platelet transfusion.
* Absolute neutrophil count (ANC) must be >500/ µl without myeloid growth factor support.
* Should not be receiving erythropoietin and/or myeloid growth factor for at least 14 days prior to initiation of study therapy.
* Should not have current diagnosis or prior history of any autoimmune or immune deficiency disorders including human immunodeficiency virus positive/acquired immunodeficiency syndrome (HIV+/AIDS).
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* Both male and female and members of all races and ethnic groups are eligible for this study.

Exclusion Criteria:

* Prior therapy with lenalidomide.
* Proliferative chronic myelomonocytic leukemia (CMML with WBC≥12,000/µL in peripheral blood), confirmed by bone marrow biopsy.
* Acute myelogenous leukemia with bone marrow myeloblast ≥30%
* MDS secondary to treatment with radiotherapy, chemotherapy, and/or immunotherapy for malignant or autoimmune diseases are excluded.
* Any of the following laboratory abnormalities:

  * Serum creatinine > 1.5 x upper limit of normal (ULN)
  * Serum aspartic transaminase (AST) or alanine transaminase (ALT) >2.0 x ULN
  * Serum total bilirubin > 2.0 mg/dL (34 µmol/L)
* Prior ≥ grade-2 national Cancer Institute Common Toxicity Criteria (NCI CTC) allergic reaction to thalidomide.
* Prior desquamating (blistering) rash while taking thalidomide.
* Prior allergic reaction to vaccination of any sort.
* Participants with ≥ grade-2 neuropathy.
* Clinically significant anemia due to factors such as iron, B12 or folate deficiencies, autoimmune or hereditary hemolysis or gastrointestinal bleeding.
* Use of cytotoxic chemotherapeutic agents, growth factors, or experimental agents (agents that are not commercially available) for the treatment of MDS within 28 days of the start of drug treatment.
* Prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix) unless the participant has been free of disease for ≥3 years.
* Any serious medical condition or psychiatric illness that will prevent the participant from signing the informed consent form or will place the participant at unacceptable risk if he/she participates in the study.
* Pregnant or nursing females.
* Use of corticosteroids greater than the equivalent of prednisone 10mg daily within 4 weeks of the first vaccination, and on-going need for corticosteroids greater than the equivalent of prednisone 10 mg daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-02-02 (Actual); Primary Completion 2014-02-17 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 24 months
  Determination of MTD of GM.CD40L bystander vaccine with lenalidomide in high-risk MDS patients.

SECONDARY OUTCOMES:
Number of Participants with Toxicities | 24 months
  Determination of toxicities associated with combination of GM.CD40L bystander vaccine with lenalidomide in high-risk MDS patients.
Number of Participants with Augmentation of Specific T Cell Immunological Functions | 24 months
  Augmentation of specific T cell immunological functions; T cell proliferation and Interferon-γ production, delayed type hypersensitivity (DTH) sensitivity by lenalidomide.
Number of Participants with Reduction of Bone Marrow Myeloblast | 24 months
  Reduction of bone marrow myeloblast from baseline to post treatment with lenalidomide and GM.CD40L bystander vaccine.
Number of Participants with Improvement of Hemoglobin and/or red blood cell (RBC) Transfusion Independence | 24 months
  Improvement of hemoglobin and/or RBC transfusion independence after combined immunotherapy treatment.
Number of Participants with Resolution of Karyotypic Changes | 24 months
  Resolution of karyotypic changes after combined treatment.
Number of Participants with Augmentation of Other T Cell Parameters | 24 months
  Augmentation of other T cell parameters after the combined treatment.
Duration of Response | 24 months
  Determination of response duration evaluated by Wilms Tumor 1 (WT1) expression and clinical outcomes. Clinical response will be assessed using International Working Group (IWG) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pinilla, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer & Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States